CLINICAL TRIAL: NCT07364318
Title: Cognitive Function and Pathophysiological Mechanisms in Adults With Obstructive Sleep Apnea: Long-term Impact of Positive Airway Pressure Therapy
Brief Title: Cognitive Function in Obstructive Sleep Apnea
Acronym: CUFM1DN
Status: Recruiting | Type: Observational
Sponsor: Comenius University (Other)
Collaborators: University Hospital Bratislava (Other); Slovak Academy of Sciences (Other Government)
Responsible Party: Sponsor
Other Study IDs: CUFM1DN-0111202431122025; VEGA 1/0075/25 (Other Grant/Funding Number: Ministry of education and science)
Record Dates: First submitted 2025-11-14; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: OSA - Obstructive Sleep Apnea; Cognitive Functions
Keywords: Cognitive Function; Positive Airway Pressure Therapy; Obstructive Sleep Apnea; Neuroimaging; Biomarkers; Vascular Changes; Metabolic Changes
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — blood and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newly diagnosed OSA: Newly diagnosed OSA according to the criteria of the American Academy of Sleep Medicine Guidelines (overnight PSG with an AHI ≥5 events per hour, hypopneas defined by ≥ 10 seconds of airflow reduction accompanied by ≥ 3% desaturation or an arousal).

SUMMARY:
Obstructive sleep apnea (OSA) is the most common sleep-related breathing disorder and has been increasingly recognized as a contributor to cognitive decline and a potential risk factor for neurodegeneration. Previous studies have identified several associated comorbidities, including vascular dysfunction, metabolic alterations, and neuroinflammatory changes. However, the impact and underlying interplay of these pathophysiological mechanisms remain poorly understood due to the lack of integrated, multidimensional assessment. This prospective, observational, longitudinal cohort study aims to investigate cognition and OSA-related physiological and pathophysiological processes in 100 adults newly diagnosed with OSA, who have no history of chronic diseases (except for overweight and obesity) and are not receiving chronic medication. A subgroup of patients with moderate to severe OSA indicated for positive airway pressure (PAP) therapy will be followed to evaluate its long-term effects on cognitive function and related mechanisms. All participants will undergo polysomnography (PSG), comprehensive neuropsychological assessment, brain MRI with volumetric analysis, biomarker profiling from blood and saliva, and evaluation of endothelial function, baroreflex sensitivity, and gut microbiome composition at baseline and after 12 months. PAP adherence will be continuously monitored. The primary objective of this study is to characterize the profile of cognitive impairment associated with OSA. Secondary exploratory analyses will focus on factors contributing to neurocognitive dysfunction in OSA.

DETAILED DESCRIPTION:
1. Background OSA is a multifaceted sleep disorder characterized by repeated episodes of upper airway obstruction during sleep, leading to significant reductions in airflow and oxygenation. Beyond its primary respiratory manifestations, OSA is associated with major comorbidities such as cardiovascular, metabolic, and neurocognitive disorders, affecting overall health and quality of life. Epidemiological data suggest that OSA affects nearly one billion individuals worldwide, yet remains markedly underdiagnosed, particularly in middle-aged and older adults. Chronic intermittent hypoxia and sleep fragmentation have been implicated in the disruption of neural networks involved in attention, executive function, memory, and emotion regulation. Neuroimaging studies further support these findings, revealing region-specific brain alterations such as hippocampal and cortical atrophy, white-matter hyperintensities, and changes in cerebral perfusion and metabolism. These mechanisms may contribute to accelerated brain aging and increase the vulnerability to neurodegenerative processes. With the global rise in dementia and aging populations, identifying modifiable contributors to cognitive decline is critical. Given that OSA is a treatable condition, timely diagnosis and effective management may represent one of the most accessible interventions to prevent or delay cognitive deterioration in vulnerable populations.
2. Aim of the study The primary aim of this study is to perform a detailed cognitive assessment in patients with OSA. The investigators seek to analyze the baseline prevalence, severity, and pattern of cognitive deficits in this population to gain a clearer understanding of the initial cognitive status from which potential therapeutic or disease-related changes may occur. The secondary aims of this study are exploratory. The investigators plan to investigate potential associations between cognitive impairment and a spectrum of PSG, sleep-related, neuroimaging, anthropometric, laboratory, and vascular measures. The investigators aim to compare the sensitivity of the Montreal Cognitive Assessment (MoCA) with that of a comprehensive neuropsychological battery. Furthermore, the investigators will evaluate the longitudinal effects of PAP therapy on cognition and the related processes under investigation.
3. Inclusion criteria Patients with newly diagnosed OSA who have no history of other chronic diseases except for overweight and obesity, are not taking any medication, and are aged between 18 and 65 years.
4. Study methodology This is a prospective, observational, single-centre cohort study conducted at the Sleep Laboratory of the 1st Department of Neurology, Faculty of Medicine, Comenius University and University Hospital Bratislava. One hundred adults with OSA will be examined at baseline and after 12 months. As part of standard clinical care, all participants will undergo overnight diagnostic PSG to confirm the OSA diagnosis and determine its severity. Patients indicated for PAP therapy will start treatment according to clinical indications, with adherence monitored via device memory cards. Additional research assessments include neuropsychological testing, brain MRI with volumetry, blood and saliva biomarker analysis, assessment of vascular functions, anthropometric measurements, oxidative stress evaluation, and gut microbiome analysis. All assessments will be performed by trained research personnel in a standardized order. Participants will first be hospitalized to undergo PSG to confirm the OSA diagnosis. After confirmation, those meeting the inclusion criteria and providing informed consent will be enrolled in the study.
5. What are the possible benefits and risks of participating? Participants may benefit from early detection of cognitive dysfunction, metabolic or vascular abnormalities, and sleep-related pathology. Risks associated with study participation are minimal and primarily related to standard blood sampling and mild discomfort during assessments. No experimental or invasive interventions are applied.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent.
2. Age 18 - 65 years.
3. Newly diagnosed OSA according to the criteria of the American Academy of Sleep Medicine Guidelines (overnight PSG with an AHI ≥5 events per hour, hypopneas defined by ≥ 10 seconds of airflow reduction accompanied by ≥ 3% desaturation or an arousal).
4. Able to accomplish relevant tests and follow-up.

Exclusion Criteria:

1. History of any chronic disease other than overweight and obesity.
2. Severe psychiatric condition that could affect cognitive functions.
3. Chronic use of medication or nicotine that may affect the study results.
4. Prior neuropsychological assessment less than 6 months before the start of the research.
5. Prior therapy for OSA (i.e., CPAP, upper airway surgery, or oral appliance).
6. Motor or sensory deficits that would significantly complicate test administration.
7. Patients who do not have Slovak as their native language actively used in daily communication.
8. Considered by the study team as not suitable for enrollment based on clinical judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed OSA who have no history of other chronic diseases except for overweight and obesity, are not taking any medication, and are aged between 18 and 65 years.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rey Auditory - Verbal Learning Test (RAVLT) | Baseline
  Measure of verbal episodic memory, encompassing immediate recall, learning across trials, delayed recall, and recognition.
  Units: total number of correctly recalled words (0-75); z-score. Higher scores indicate better performance.
Figure Copy Task | Baseline
  A visuoconstructional task used to assess visual perception, spatial planning, and visual memory.
  Units: score 0-24 points; z-score. Higher scores indicate better performance.
Controlled Oral Word Association Test (COWAT) | Baseline
  A verbal fluency task requiring rapid generation of words beginning with specified letters. It assesses phonemic fluency, executive function, and lexical retrieval.
  Units: number of correct words generated per minute; z-score. Higher scores indicate better performance.
Category Fluency Test | Baseline
  A semantic fluency measure where subjects list as many words from a given category. It evaluates semantic memory and executive retrieval processes.
  Units: number of correct words generated per minute; z-score. Higher scores indicate better performance.
Trail Making Test (TMT) | Baseline
  A two-part test evaluating processing speed, visual search, attention, and task-switching.
  Units: completion time in seconds; z-score. Shorter completion times indicate better performance.
The Stroop Color and Word Test | Baseline
  Measure of selective attention, processing speed, cognitive flexibility, and inhibitory control.
  Units: completion time in seconds; z-score. Shorter completion times indicate better performance.
Digit Span | Baseline
  A working memory test comprising forward and backward recall of digit sequences. Assesses attention, concentration, and short-term memory.
  Units: total score (0-14 points); z-score. Higher scores indicate better performance.
Montreal Cognitive Assessment (MoCA) | Baseline
  General cognition screening targeting attention, executive function, memory, language, visuospatial abilities, and orientation.
  Units: total score (0-30 points); ≥26 = normal cognition. Higher scores indicate better performance.
Generalized Anxiety Disorder 7-item scale (GAD - 7) | Baseline
  A 7-item self-report questionnaire to screen and assess the severity of generalized anxiety disorder. Items are rated on a 4-point scale. Units: total score (0-21 points); cut-off ≥ 10. Higher scores indicate greater anxiety symptom severity.
Patient´s Health Questionnaire (PHQ - 9) | Baseline
  A 9-item scale assessing depression severity based on DSM IV criteria. Items are rated on a 4-point scale.
  Units: total score (0-27 points); cut-off ≥ 10. Higher scores indicate greater depressive symptom severity.
Rey Auditory - Verbal Learning Test (RAVLT) 12 moths | Change from baseline to 12 months
  Measure of verbal episodic memory, encompassing immediate recall, learning across trials, delayed recall, and recognition.
  Units: total number of correctly recalled words (0-75); z-score. Higher scores indicate better performance. Assessments will be performed after 12 months.
Figure Copy Task 12 months | Change from baseline to 12 months
  A visuoconstructional task used to assess visual perception, spatial planning, and visual memory.
  Units: score 0-24 points; z-score. Higher scores indicate better performance. Assessments will be performed after 12 months.
Controlled Oral Word Association Test (COWAT) 12 months | Change from baseline to 12 months
  A verbal fluency task requiring rapid generation of words beginning with specified letters. It assesses phonemic fluency, executive function, and lexical retrieval.
  Units: number of correct words generated per minute; z-score. Higher scores indicate better performance. Assessments will be performed after 12 months.
Category Fluency Test 12 months | Change from baseline to 12 months
  A semantic fluency measure where subjects list as many words from a given category. It evaluates semantic memory and executive retrieval processes.
  Units: number of correct words generated per minute; z-score. Higher scores indicate better performance.
  Assessments will be performed after 12 months.
Trail Making Test (TMT) 12 months. | Change from baseline to 12 months
  A two-part test evaluating processing speed, visual search, attention, and task-switching.
  Units: completion time in seconds; z-score. Shorter completion times indicate better performance.
  Assessments will be performed after 12 months.
The Stroop Color and Word Test 12 months. | Change from baseline to 12 months
  Measure of selective attention, processing speed, cognitive flexibility, and inhibitory control.
  Units: completion time in seconds; z-score. Shorter completion times indicate better performance.
  Assessments will be performed after 12 months.
Digit Span 12 months. | Change from baseline to 12 months
  A working memory test comprising forward and backward recall of digit sequences. Assesses attention, concentration, and short-term memory.
  Units: total score (0-14 points); z-score. Higher scores indicate better performance.
  Assessments will be performed after 12 months.
Montreal Cognitive Assessment (MoCA) 12 months. | Change from baseline to 12 months
  General cognition screening targeting attention, executive function, memory, language, visuospatial abilities, and orientation.
  Units: total score (0-30 points); ≥26 = normal cognition. Higher scores indicate better performance.
  Assessments will be performed after 12 months.
Generalized Anxiety Disorder 7-item scale (GAD - 7) 12 months. | Change from baseline to 12 months
  A 7-item self-report questionnaire to screen and assess the severity of generalized anxiety disorder. Items are rated on a 4-point scale. Units: total score (0-21 points); cut-off ≥ 10. Higher scores indicate greater anxiety symptom severity.
  Assessments will be performed after 12 months.
Patient´s Health Questionnaire (PHQ - 9) 12 months. | Change from baseline to 12 months
  A 9-item scale assessing depression severity based on DSM IV criteria. Items are rated on a 4-point scale.
  Units: total score (0-27 points); cut-off ≥ 10. Higher scores indicate greater depressive symptom severity.
  Assessments will be performed after 12 months.

SECONDARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | Baseline
  A polysomnographic measure representing the number of apneas and hypopneas per hour of sleep.
  Units: events per hour. Higher scores indicate more severe OSA.
Apnea-Hypopnea Index (AHI) 12 months | 12 months
  A polysomnographic measure representing the number of apneas and hypopneas per hour of sleep.
  Units: events per hour. Higher scores indicate more severe OSA. Assessments will be performed after 12 months.
Positive Airway Pressure (PAP) Therapy Adherence | 12 months
  Objective measure of treatment compliance obtained from PAP device data. Units: average hours of use per night. Higher scores indicate better adherence to therapy. Assessments will be performed after 12 months.
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline to 12 months
  A self-rated questionnaire comprising 19 items that evaluate sleep quality and disturbances over a one-month interval.
  Units: global PSQI score (0-21 points); cut-off ≥ 5. Higher scores indicate poorer overall sleep quality.
Epworth Sleepiness Scale (ESS) | Change from baseline to 12 months
  An 8-item self-report questionnaire measuring habitual daytime sleepiness in common situations.
  Units: total score (0-24 points); cut-off ≥ 10. Higher scores indicate greater daytime sleepiness.
Brain Volumetry | Change from baseline to 12 months
  Quantitative assessment of total and regional brain volumes will include total brain volume, gray and white matter volumes, hippocampal volume, cortical thickness, and other regional volumetric measures.
  Units: mL; changes in volumes reflect structural brain alterations.
Body Mass Index (BMI) | Change from baseline to 12 months
  BMI calculated as weight (kg) divided by height squared (m²). Units: kg/m². Higher values indicate greater adiposity.
Apolipoprotein E (APOE) | Baseline
  Genotype Genetic biomarker associated with neurodegenerative risk. Units: genotype category (ε2/ε2, ε2/ε3, ε2/ε4, ε3/ε3, ε3/ε4, ε4/ε4). ε4 allele presence indicates higher vulnerability to cognitive decline.
Plasma Neurofilament Light Chain (pNfL) | Change from baseline to 12 months
  A biomarker of neuroaxonal injury. Units: pg/mL. Higher concentrations indicate greater neuronal damage.
Total cholesterol | Change from baseline to 12 months
  Measure of circulating total cholesterol, representing the combined cholesterol content within all lipoprotein classes.
  Units: mmol/L. Higher values reflect a more adverse lipid profile.
Trolox Equivalent Antioxidant Capacity (TEAC) | Change from baseline to 12 months
  Measure of total antioxidant capacity in plasma and saliva. Units: mmol Trolox equivalents/L. Lower TEAC values indicate reduced antioxidant defense and increased susceptibility to oxidative stress.
Reactive Hyperemia Index (RHI) | Change from baseline to 12 months
  Measure of endothelial function assessed by pulse amplitude tonometry. RHI reflects the vasodilatory response of peripheral arteries following temporary occlusion.
  Units: ratio. Lower values indicate worse endothelial function.
Baroreflex Sensitivity | Change from baseline to 12 months
  Indicator of autonomic cardiovascular regulation measured via Finometer. Units: ms/mmHg. Higher values indicate better baroreflex control.
Gut Microbiome Composition | Change from baseline to 12 months
  Analysis of microbial diversity and abundance from stool samples. Units: Shannon index and Bray-Curtis dissimilarity. Lower alpha diversity and altered beta diversity indicate dysbiosis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Turcani, prof. MD PhD., Study Director — 1st Department of Neurology, Faculty of Medicine, Comenius University and University Hospital Bratislava, Slovakia
Locations (1):
- 1st Department of Neurology, Faculty of Medicine, Comenius University and University Hospital Bratislava, Slovakia, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No
The study results will present the group as a whole, not individual patient data.

REFERENCES:
- [Result] Sehr T, Akgun K, Benkert P, Kuhle J, Ziemssen T, Brandt MD. Effects of obstructive sleep apnea treatment on neurodegenerative biomarker neurofilament light chain and cognitive performance. J Sleep Res. 2024 Oct;33(5):e14164. doi: 10.1111/jsr.14164. Epub 2024 Feb 13. PMID 38351662
- [Result] Xue X, Zhao Z, Zhao LB, Gao YH, Xu WH, Cai WM, Chen SH, Li TJ, Nie TY, Rui D, Ma Y, Qian XS, Lin JL, Liu L. Gut microbiota changes in healthy individuals, obstructive sleep apnea patients, and patients treated using continuous positive airway pressure: a whole-genome metagenomic analysis. Sleep Breath. 2024 Nov 26;29(1):11. doi: 10.1007/s11325-024-03185-z. PMID 39589660
- [Result] Silva WA, Almeida-Pititto B, Santos RB, Aielo AN, Giatti S, Parise BK, Souza SP, Vivolo SF, Lotufo PA, Bensenor IM, Drager LF. Obstructive sleep apnea is associated with lower adiponectin and higher cholesterol levels independently of traditional factors and other sleep disorders in middle-aged adults: the ELSA-Brasil cohort. Sleep Breath. 2021 Dec;25(4):1935-1944. doi: 10.1007/s11325-021-02290-7. Epub 2021 Feb 15. PMID 33590375
- [Result] Salari N, Khazaie H, Abolfathi M, Ghasemi H, Shabani S, Rasoulpoor S, Mohammadi M, Rasoulpoor S, Khaledi-Paveh B. The effect of obstructive sleep apnea on the increased risk of cardiovascular disease: a systematic review and meta-analysis. Neurol Sci. 2022 Jan;43(1):219-231. doi: 10.1007/s10072-021-05765-3. Epub 2021 Nov 19. PMID 34797460
- [Result] Durtette A, Dargent B, Gierski F, Barbe C, Deslee G, Perotin JM, Henry A, Launois C. Impact of continuous positive airway pressure on cognitive functions in adult patients with obstructive sleep apnea: A systematic review and meta-analysis. Sleep Med. 2024 Nov;123:7-21. doi: 10.1016/j.sleep.2024.08.019. Epub 2024 Aug 22. PMID 39226674
- [Result] Bubu OM, Andrade AG, Umasabor-Bubu OQ, Hogan MM, Turner AD, de Leon MJ, Ogedegbe G, Ayappa I, Jean-Louis G G, Jackson ML, Varga AW, Osorio RS. Obstructive sleep apnea, cognition and Alzheimer's disease: A systematic review integrating three decades of multidisciplinary research. Sleep Med Rev. 2020 Apr;50:101250. doi: 10.1016/j.smrv.2019.101250. Epub 2019 Dec 12. PMID 31881487
- [Result] Xu H, Liu Y, Li C, Li X, Shen L, Wang H, Liu F, Zou J, Xia Y, Huang W, Liu Y, Gao Z, Fu Y, Wang F, Huang S, Song Z, Song F, Gao Y, Peng Y, Zou J, Zhu H, Liu S, Li L, Zhu X, Xiong Y, Hu Y, Yang J, Li Y, Gao F, Guo Q, Huang H, Zhang W, Li J, Chen Y, Dong P, Yang J, Lv J, Wang P, Sun Y, Qian B, Yaffe K, Guan J, Yi H, Leng Y, Yin S. Effects of Continuous Positive Airway Pressure on Neuroimaging Biomarkers and Cognition in Adult Obstructive Sleep Apnea: A Randomized Controlled Trial. Am J Respir Crit Care Med. 2025 Apr;211(4):628-636. doi: 10.1164/rccm.202406-1170OC. PMID 39998447